CLINICAL TRIAL: NCT02217865
Title: Patient-Centered Risk Adjusted Surveillance After Curative Resection of Colorectal Cancer
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); Alliance for Clinical Trials in Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: PA13-1002; CE13-04-6855 (Other Grant/Funding Number: Patient-Centered Outcomes Research Institute); NCT02321488 (obsolete NCT alias)
Record Dates: First submitted 2014-08-13; First posted 2014-08-15 (Estimated); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Colorectal Cancer
Keywords: Colorectal Cancer; CRC; Curative resection of colorectal cancer; Caregivers; Interviews; Focus groups; Questionnaires; Surveys
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Surveys and Questionnaires; Focus Groups

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

GROUPS / COHORTS (2):
- Colorectal Cancer Participants: Colorectal cancer participants undergoing follow-up after curative resection of colorectal cancer.
  Interventions: Behavioral: Interviews - Colorectal Cancer Participants; Behavioral: Questionnaire; Behavioral: Focus Groups
- Caregivers of Colorectal Cancer Participants: Caregivers of colorectal cancer participants undergoing follow-up after curative resection of colorectal cancer.
  Interventions: Behavioral: Interviews - Colorectal Cancer Participants; Behavioral: Focus Groups; Behavioral: Interviews - Caregivers of Colorectal Cancer Participants

INTERVENTIONS:
Behavioral: Interviews - Colorectal Cancer Participants — Semi-structured interviews conducted exploring key issues relevant to colorectal cancer surveillance following curative resection. Interviews take between 30 minutes and 1 hour.
Behavioral: Questionnaire — Questionnaire completion asking general health and demographic questions.
  Other Names: Survey
  Groups: Colorectal Cancer Participants
Behavioral: Focus Groups — Focus groups conducted with participants and caregivers. Up to 4 focus groups conducted with up to 30 participants each. Focus groups expected to take 30 to 60 minutes.
Behavioral: Interviews - Caregivers of Colorectal Cancer Participants — Semi-structured interviews conducted exploring key issues relevant to colorectal cancer surveillance following curative resection. Interviews take between 30 minutes and 1 hour.
  Groups: Caregivers of Colorectal Cancer Participants

SUMMARY:
The long-term goal of this research is to develop new tools to guide patients, caregivers, and clinicians in making individualized decisions regarding colorectal cancer (CRC) surveillance. As part of a Patient-Centered Outcomes Research Institute-funded contract, investigator will analyze surveillance data to determine the effectiveness of CRC surveillance and recurrence risk taking into account different patient and tumor characteristics; identify key issues about CRC surveillance important to patients, caregivers, and clinicians; and integrate the recurrence risk and patient priorities into a patient-centered, risk stratified surveillance strategy by creating an interactive decision aid for use by patients and clinicians.

This protocol addresses a formative step in the creation of the interactive decision aid where patients' information needs and preferences are assessed regarding decisions about surveillance.

The specific aims of this protocol are:

Phase 1 - To interview patients and their caregivers to determine their concerns, preferences and key priorities regarding surveillance after curative resection of colorectal cancer, and

Phase 2 - To refine the key priorities identified in phase 1 through focus groups and surveys with patients and caregivers.

DETAILED DESCRIPTION:
You are being asked to take part in this research study which is conducted at The University of Texas MD Anderson ("MD Anderson") and the Harris Health System because you (or someone you act as a caregiver for) are undergoing follow-up after curative resection of colorectal cancer.

The goal of this study is to find out the key priorities for patients and their caregivers when it comes to surveillance after curative resection of colorectal cancer. Your responses will help develop decision aids to help future colorectal cancer patients make more informed decisions about surveillance.

If you agree to participate in this study, you will take part in an interview or focus group in person at MD Anderson, the Harris Health System, or the Alliance. The interview or focus group is expected to take between 30 minutes and 1 hour. The interview or focus group will be audiorecorded. Your name or other identifying information will not appear in the transcript. Adept Word Management, a transcription service that has been approved by the institution, may transcribe the interviews.

You will be asked questions about:

* your priorities and concerns about colorectal cancer surveillance
* what you know about colorectal cancer and surveillance,
* your cancer and treatment (or the patients'),
* the impact or inconvenience that surveillance causes,
* who you think should make decisions about surveillance,
* your thoughts about different surveillance scenarios,
* and general questions about your age, race, sex, education, and income level.

Information about you will be collected from the medical records and existing data in a database of colorectal patients that is used to organize existing information about colorectal patients to better understand the disease. Information collected will include things like age, gender, marital status, information about the tumor, type of surgery, and what treatment was done before and after surgery. There are no other plans to share your information with others outside the study.

Your participation will be over when the interview is complete. If you are undergoing follow-up for colorectal cancer, research staff will look at your medical record after the interview for information about your cancer including tumor characteristics.

Your participation is completely voluntary. Whether you say yes or no will not change your medical care.

Up to 220 patients and their caregivers will participate in this multicenter study. Up to 190 patients and their caregivers will be enrolled at MD Anderson. Up to 10 patients and their caregivers will be enrolled at the Harris Health System.

ELIGIBILITY:
Inclusion Criteria:

1. Age 21 or older
2. Able to read and speak English
3. Able to undergo a 30 to 60-minute interview or focus group
4. For phase 1: MD Anderson patient undergoing follow-up for curative resection of stage I-IV colon or rectal cancer OR caregiver of such a patient
5. For phase 2: Colon or rectal cancer patient

Exclusion Criteria:

N/A

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients of MD Anderson Colorectal Center and their caregivers recruited by study staff.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2014-07-16 (Actual); Primary Completion 2022-01-13 (Actual); Study Completion 2022-01-13 (Actual)

PRIMARY OUTCOMES:
Effectiveness of Colorectal Cancer (CRC) Surveillance | 1 day
  Semi-structured interviews and focus groups reviewed to identify themes related to participants' and caregiver's priorities regarding surveillance of colorectal cancer.

CONTACTS AND LOCATIONS:
Overall Officials: George J. Chang, MD,MS, Study Chair — M.D. Anderson Cancer Center; Robert Volk, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (3):
- United States (3):
  - University of California San Francisco, San Francisco, California
  - Lyndon B. Johnson General Hospital, Houston, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Zafar SN, Hu CY, Snyder RA, Cuddy A, You YN, Lowenstein LM, Volk RJ, Chang GJ. Predicting Risk of Recurrence After Colorectal Cancer Surgery in the United States: An Analysis of a Special Commission on Cancer National Study. Ann Surg Oncol. 2020 Aug;27(8):2740-2749. doi: 10.1245/s10434-020-08238-7. Epub 2020 Feb 20. PMID 32080809
- [Derived] Snyder RA, Hu CY, Cuddy A, Francescatti AB, Schumacher JR, Van Loon K, You YN, Kozower BD, Greenberg CC, Schrag D, Venook A, McKellar D, Winchester DP, Chang GJ; Alliance for Clinical Trials in Oncology Network Cancer Surveillance Optimization Working Group. Association Between Intensity of Posttreatment Surveillance Testing and Detection of Recurrence in Patients With Colorectal Cancer. JAMA. 2018 May 22;319(20):2104-2115. doi: 10.1001/jama.2018.5816. PMID 29800181
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org